CLINICAL TRIAL: NCT03632018
Title: Heart Exercise And Resistance Training - Peer Lead ActivitY (HEART-PLAY)
Brief Title: Heart Exercise And Resistance Training - Peer Lead ActivitY
Acronym: HEART-PLAY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Paul J. Mills, Professor IR, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01HL136407 (NIH)
Record Dates: First submitted 2018-07-30; First posted 2018-08-15 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular Diseases
Keywords: cardiac rehabilitation; physical activity
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Because we are intentionally changing the clinic environment, study participants and care providers will not be masked to the study condition. However, the investigator and the outcome assessors will be unaware which study arm a given participant is in to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Cardiac Rehabilitation (Active Comparator): Participants in the STANDARD condition will receive the standard of care cardiac rehabilitation, consisting of 36 sessions across 12 weeks of prescribed, supervised exercise sessions.
  Interventions: Behavioral: Standard Cardiac Rehabilitation
- HEART-PLAY (Experimental): Participants in the HEART-PLAY will receive standard CR and additionally receive pedometers, resistance bands, and the National Institute of Aging (NIA) exercise guide. They will further receive counseling from peer health coaches, social support from group education sessions, and supplemental educational materials. After the 12 weeks of prescribed, supervised exercise sessions, HEART-PLAY group participants will continue to receive support from peers and clinic staff with check-in calls, feedback on pedometer goals, and twice weekly group events including walks and/or resistance band group exercise classes.
  Interventions: Behavioral: HEART-PLAY

INTERVENTIONS:
Behavioral: HEART-PLAY — Participants assigned to the HEART-PLAY intervention will receive standard CR. Additionally, they will receive pedometers, group education, and educational materials introduced by peer Health Coaches for 12 months. Before or after their regularly scheduled CR appointments, they will meet at the clinic as a group twice per week to receive Health Tips and participate in discussions. At 8 weeks in to the 12-week CR, they will begin to discuss with their peer Health Coaches the transition from the formal CR setting into community-based exercise. As part of this transition, peer Health Coaches will slowly introduce group community walks and train participants in the proper use of resistance bands. Health Coaches will have talk with their assigned participants about relapse prevention and sustaining exercise following the termination of formal CR.
  Arms: HEART-PLAY
Behavioral: Standard Cardiac Rehabilitation — During the 12-week intervention period, the STANDARD intervention participants will receive standard of care by attending the 36 sessions of standard CR as prescribed by his/her physician and administered by the Step Clinic.
  Arms: Standard Cardiac Rehabilitation

SUMMARY:
Numerous studies show that regular physical activity / exercise significantly improves exercise tolerance as well as clinical outcomes in cardiovascular disease (CVD). Exercise as a reliable adjunctive intervention, however, remains limited due to poor short- as well as long-term adherence. The study examines the effectiveness of the peer-led Heart Exercise And Resistance Training - Peer Lead ActivitY (HEART-PLAY) intervention to significantly sustain exercise adherence among CR patients, as compared a standard CR intervention. In a rigorous cluster randomized controlled trial at the UCSD Step Family Cardiovascular Rehabilitation and Wellness Center, the study assesses the HEART-PLAY intervention program in 264 socioeconomically and ethnically diverse women and men 18+ years old who have been referred to standard CR. Participants in the HEART-PLAY and in the STANDARD CR programs will both participate in 36 sessions of CR across approximately 12 weeks, as prescribed by their physician. Participants in HEART-PLAY will additionally receive peer and staff leadership, self-monitoring tools and feedback, group education and materials, and motivational, goal-setting, and relapse prevention counseling sessions. The study will demonstrate that the peer-led HEART-PLAY program based in the clinic setting will significantly enhance the primary study endpoint of adherence to 150 min/week of moderate physical activity/week.

DETAILED DESCRIPTION:
This study examines the effectiveness of the Heart Exercise And Resistance Training - Peer Lead ActivitY (HEART-PLAY) intervention to significantly sustain exercise adherence in patients referred for Cardiac Rehabilitation (CR). CR Clinic staff and CR patients who meet study inclusion criteria and are willing to serve as peer leaders, will be taught to lead the intervention activities with trained health educators and research staff. The HEART-PLAY program and behavior change will be sustainable because of the presence of peer and staff leadership and because it employs proven strategies from social cognitive theory and ecological models including self-monitoring, feedback, social support, role modeling, and relapse prevention. HEART-PLAY teaches patients how to accumulate meaningful PA across the day and provides a supportive social infrastructure to maintain motivation. Since the aim is to test an augmented CR program that can be widely adopted, the project employs a design that allows for the concurrent testing of both intervention and implementation strategies and outcomes. Across the five days of the week and the AM and PM clinic sessions, there will be approximately 25 different peer-led groups (clusters) run to obtain complete data on a total of 264 women and men 18+ years old of varied socioeconomic and ethnic backgrounds referred for CR. HEART-PLAY and STANDARD participants will be scheduled to visit the Step Clinic on distinctly different days/times to avoid contamination. Participants in the STANDARD condition will receive the standard of care cardiac rehabilitation, consisting of 36 sessions across 12 weeks of prescribed, supervised exercise sessions, Participants in the HEART-PLAY will receive standard CR and additionally receive pedometers, resistance bands, and the National Institute of Aging (NIA) exercise guide. Patients will further receive counseling from peer health coaches, social support from group education sessions, and supplemental educational materials. After the 12 weeks of prescribed, supervised exercise sessions, HEART-PLAY group participants will continue to receive support from peers and clinic staff with check-in calls, feedback on pedometer goals, and bi-weekly group events including walks and/or resistance band group exercise classes. Pilot data support that the peer-led approach in the clinic setting will be enthusiastically received by patients and significantly increase PA and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Referred to the UCSD Step Clinic for 36 sessions of cardiac rehabilitation across 12-14 weeks for one of the following medical conditions: myocardial infarction, coronary artery bypass surgery, stable angina, heart valve repair or replacement, coronary angioplasty or stenting, or congestive heart failure.
* Able to give informed consent in English
* Able to perform study assessments as described
* Blood pressure <180/110 mmHg
* Able to perform light to moderate exercise
* Have not had a fall during the previous 6 months resulting in an injury
* Clinical staff's permission to participate, including their assessment that participant is a good candidate for this particular research study
* Ability to complete written or computer-based surveys
* Completion of a post-consent comprehension test

Exclusion Criteria:

* Referred to CR following VAD (Ventricular Assist Device) procedure, peripheral arterial disease (PAD), or heart or lung transplant. Angina not adequately managed with nitrates
* Oxygen-dependent COPD
* Recent stroke or significant cerebral neurologic impairment that would interfere with participation
* Major depressive disorder per eMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Minutes of Moderate Physical Activity (PA) | 3 months, 6 months, and 12 months
  7-day actigraphy records will be used to assess amount of moderate PA

SECONDARY OUTCOMES:
Change in Health-related quality of life (QoL) | 3 months, 6 months, and 12 months
  Demonstrate improved QoL as determined by the NIH-supported PROMIS-29
Improved Cost-effectiveness | 12 months
  Determine cost-effectiveness using Markov Models
Change in BNP levels | 3 months, 6 months, and 12 months
  Assess reductions in circulating cardiac health biomarkers using standard biomarkers assays
Change in Galectin-3 levels | 3 months, 6 months, and 12 months
  Assess reductions in circulating cardiac health biomarkers using standard biomarkers assays

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No